CLINICAL TRIAL: NCT06296043
Title: The Effect of Su-Jok Application and Progressive Muscle Relaxation Exercises in Coping With Premenstrual Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBU-FUT-01
Record Dates: First submitted 2024-02-12; First posted 2024-03-06 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-02

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Nursing; Su-Jok; Progressive muscle relaxation exercise
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Three groups with su-jok group, progressive muscle relaxation exercise group and control group
Who Masked: Participant
Masking Description: Double (Participant, Outcomes Assessor) Since the application will be performed by the researcher, participant will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive Muscle Relaxation Exercise Group (Experimental): Application will be made on the day PMS symptoms begin and throughout the menstrual cycle.
  Interventions: Procedure: Progressive Muscle Relaxation Exercise Group
- Su-Jok Group (Experimental): Application will be made on the day PMS symptoms begin and throughout the menstrual cycle.
  Interventions: Procedure: Su-Jok Intervention
- Control Group (No Intervention): No application will be made to this group by the researcher.

INTERVENTIONS:
Procedure: Progressive Muscle Relaxation Exercise Group — Exercise Group
  Arms: Progressive Muscle Relaxation Exercise Group
Procedure: Su-Jok Intervention — Hand massage with seeds
  Arms: Su-Jok Group

SUMMARY:
The aim of this study is to determine the effect of su-jok application and progressive muscle relaxation exercise in coping with premenstrual syndrome.

DETAILED DESCRIPTION:
Various medications can be used to relieve PMS symptoms, but there is no treatment to completely eliminate it. For this reason, women may seek traditional and alternative practices to reduce PMS complaints. Alternative methods such as herbal treatment, aromatherapy, acupuncture, nutrition regulation and stress control can be used to relieve PMS symptoms. It has been stated that applying mind-body based therapies to relieve PMS symptoms is safe and cost-effective. Such interventions include progressive muscle relaxation exercise (PCGE), paced breathing, clinical hypnosis, yoga, mindfulness, reflexology, and cognitive behavioral therapies. Su-Jok application, which is an alternative method, can also be used to relieve PMS symptoms. In Su-Jok therapy, the practitioner stimulates points on the hands and feet to activate auto-regulatory mechanisms and bring the body to a healthy state. Due to the negative effects of PMS on daily life, knowing the frequency of occurrence and risk factors is expected to contribute and guide individuals in coping with PMS. While PMS threatens the health of the individual in particular, it generally brings socio-economic burdens to the individual, family and society.

ELIGIBILITY:
Inclusion Criteria:

* Getting over 104 points from the PMS scale,
* Having regular menstruation,
* Not having any chronic disease,
* Not using any method to cope with PMS.

Exclusion Criteria:

* Having irregular menstruation,
* Having musculoskeletal system and respiratory diseases,
* Having a diagnosed psychiatric disease,
* Having a disease that may cause premenstrual symptoms and receiving medical treatment (thyroid diseases, heart failure, neurological disorders)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since it is a study conducted on premenstrual symptoms with women, it concerns the female gender.
Enrollment: 135 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
PAIN Visual Analog Scale (VAS)- (Min:0 - Max:10) | 3 months
  In the 1st, 2nd and 3rd month menstrual periods;
  * Premenstrual Syndrome Scale
  * VAS evaluation scale will be applied.
FATIGUE Visual Analog Scale (VAS)- (Min:0 - Max:10) | 3 months
  In the 1st, 2nd and 3rd month menstrual periods;
  * Premenstrual Syndrome Scale
  * VAS evaluation scale will be applied.
SLEEP STATE Visual Analog Scale (VAS)- (Min:0 - Max:10) | 3 months
  In the 1st, 2nd and 3rd month menstrual periods;
  * Premenstrual Syndrome Scale
  * VAS evaluation scale will be applied.
NAUSEA VOMITING Visual Analog Scale (VAS)- (Min:0 - Max:10) | 3 months
  In the 1st, 2nd and 3rd month menstrual periods;
  * Premenstrual Syndrome Scale
  * VAS evaluation scale will be applied.
Change in Premenstrual Symptoms (People with PMS scale scores over 104 points will be determined). | 3 months
  In the 1st, 2nd and 3rd month menstrual periods;
  * Premenstrual Syndrome Scale
  * VAS evaluation scale will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Ünal Toprak, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Sevil Albayrak, PhD, Principal Investigator — Kıbrıs İlim Üniversitesi
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No